CLINICAL TRIAL: NCT06002308
Title: Influence of Injury to the Kaplan Fibers and Anterolateral Ligament on Anterolateral Rotatory Knee Laxity in Adult and Pediatric Patients With Anterior Cruciate Ligament Injury: A Retrospective Cohort Study
Brief Title: Influence of Injury to the Kaplan Fibers in Adult and Pediatric Patients With ACL Injury
Status: Completed | Type: Observational
Sponsor: Sichuan Province Orthopetic Hospital (Other)
Responsible Party: Principal Investigator, Jiaming Cui, Attending Doctor, Sichuan Province Orthopetic Hospital
Other Study IDs: KY2023-018-01
Record Dates: First submitted 2023-08-05; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: ACL-injury
Keywords: Rotatory instability; Kaplan fiber injury; Anterolateral ligament; Meniscal injury; Magnetic resonance imaging; Anterior cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Age — The retrospective study included 540 patients with primary ACL tears (71 pediatric patients and 469 adults) whose MRI examination and pivot-shift test were conducted within 14 days after injury. To detect concomitant KF and ALL injury in knees with ACL injury using MRI in both adult and pediatric patients and compare the effect of KF injury and multiple risk factors on anterolateral rotatory laxity as measured by the pivot-shift test in a clinical setting.

SUMMARY:
The goal of this [type of study: observational study] is to [detect concomitant KF and ALL injury in knees with ACL injury using MRI in both adult and pediatric patients and compare the effect of KF injury and multiple risk factors (concomitant injury to the ALL, medial collateral ligament [MCL], or anterior, central, or posterior part of the medial or lateral meniscus) on anterolateral rotatory laxity as measured by the pivot-shift test in a clinical setting.].

The main question [s] it aims to answer are:

[Does the main risk factor for a high-grade pivot shift after acute ACL injury differ between pediatric patients and adults?] [Does Concomitant KF injury significantly affect the pivot-shift phenomenon in pediatric patients with acute ACL injury?] Researchers will compare [71 pediatric patients and 469 adults] to see if [main risk factor for a high-grade pivot shift after acute ACL injury differs between pediatric patients and adults?].

ELIGIBILITY:
Inclusion Criteria:

* unilateral acute primary ACL tear, considered when the patient reported knee injury occurring less than 2 weeks before the examination;
* bone bruising on the femoral condyles and tibial plateau identiﬁed on MRI.

Exclusion Criteria:

* concomitant ligament (posterior cruciate ligament and/or posterolateral complex) procedures or realignment procedures; contralateral knee injury;
* previous injury or surgery affecting the ipsilateral knee;
* insufficient data from the electronic medical record system;
* lack of KF visualization on MRI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1994 patients were identified from medical records between Jan. 2019 and Dec. 2021. After reviewing the inclusion and exclusion criteria, 540 patients were included in the present study (71 pediatric patients and 469 adults).
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
KF injury | 3 years
  concomitant KF injury or not
ALL injury | 3 years
  concomitant ALL injury or not
MCL injury | 3 years
  concomitant MCL injury or not
Medial meniscus injury | 3 years
  concomitant anterior, central, or posterior part of medial meniscus injury or not
Lateral meniscus | 3 years
  concomitant anterior, central, or posterior part of lateral meniscus injury or not

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial Orthopedic Hospital, Chengdu, Sichuan, China